CLINICAL TRIAL: NCT00438607
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Study of Single and Multiple Oral Dose Administration of BIIB014 in Subjects With Moderate to Late Stage Parkinson's Disease Who Are Also Receiving Treatment With Levodopa
Brief Title: Dose-Finding Safety Study of BIIB014 in Combination With Levodopa in Moderate to Late Stage Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 204PD202; EUDRA CT NO: 2006-003490-27; ISCRTN 12870393
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2009-07-13 (Estimated); Status verified 2009-07

CONDITIONS: Parkinson's Disease
Keywords: Moderate to late stage Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — 3-(4-amino-3-methylbenzyl)-7-(2-furyl)-3H-(1,2,3)triazolo(4,5-d)pyrimidine-5-amine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Other): BIIB014 at MTD from Part A
  Interventions: Drug: BIIB014
- 2 (Other): BIIB014 at dose immediately below MTD from Part A
  Interventions: Drug: BIIB014
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIB014 — oral administration of BIIB014 at dose to be specified from Part A, given daily for 8 weeks
  Arms: 1; 2
Drug: Placebo — Matched placebo for MTD or MTD-1
  Arms: 3

SUMMARY:
The main purpose of this study is to determine the safety of BIIB014 and how well BIIB014 is tolerated when given at different doses to patients with moderate to late-stage Parkinson's Disease who are also taking the Parkinson's medication, levodopa (L-DOPA).

This study will also explore:

1. the pharmacokinetics of BIIB014 in Parkinson's patients who are also taking L-DOPA (this will be done by measuring the levels of BIIB014 in the blood at several different times during the study), and
2. the activity of BIIB014 when given to Parkinson's patients who are also taking L-DOPA (this will be done by performing different Parkinson's Disease assessments during the study to examine change in waking OFF time, change in time with troublesome dyskinesia, change in Unified PD Rating Scale (UPDRS) scores, and Clinical Global Improvement).

Patients who enter this study will be randomly assigned to receive either BIIB014 or a placebo but because the study is blinded, neither they nor their study doctor will know which study treatment they are taking.

The study will be divided into 2 parts:

* Part A: a, rapid, sequential cohort, dose escalation to establish MTD, followed by
* Part B: a parallel-group exploration of the two highest tolerated doses versus placebo.

Note: As Part A of the study is now concluded, some of the study design information presented below (e.g., number of study arms) pertains only to Part B.

ELIGIBILITY:
Inclusion Criteria:

* Must carry a diagnosis of idiopathic PD according to UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria, and be Hoehn & Yahr Stage II to IV (inclusive) when OFF.
* Must be on a stable dose of L-3,4-dihydroxyphenylalanine (L-DOPA)/carbidopa or L-DOPA/benserazide for at least 4 weeks prior to enrollment.
* Except for L-DOPA and certain allowed dopamine agonists, must not be receiving any other PD medications. (Current treatment with certain dopamine agonists is allowed but subjects must have been on a stable dose for at least 4 weeks prior to enrollment).
* Some subjects must demonstrate a definite end of L-DOPA dose wearing off (at least 2 hours OFF time per waking day) and must be able to keep accurate patient diaries of PD activity.

Major Exclusion Criteria:

* A Mini Mental State Examination (MMSE) score <26.
* History or clinical features consistent with an atypical parkinsonian syndrome.
* Any significant non-Parkinson's central nervous system disorder.
* Any significant AXIS I psychiatric disease from the Diagnostic and Statistical Manual of Mental Disorders (DSM).
* Any previous surgical intervention for Parkinson's Disease.
* History of certain malignancies.
* History of severe allergic anaphylactic reactions to any drug.
* Clinically significant baseline electrocardiogram (ECG).
* Orthostatic hypotension.
* HbA1c >7.0%

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2007-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Number and proportion of subjects with adverse events | up to end of study
Assessment of clinical laboratory parameters | up to end of study
Assessment of vital signs | up to end of study
Assessment of ECG parameters. | up to end of study

SECONDARY OUTCOMES:
Assess PK by measuring concentrations of BIIB014 and its N-acetyl metabolite in blood plasma. | up to 24h following last dose (Part A only)
Explore activity of BIIB014 by evaluating standard Parkinson's disease assessments | up to 8h following last dose (Part A); up to 24h following last dose (Part B only)

CONTACTS AND LOCATIONS:
Overall Officials: Biogen Idec, Study Director — Cambridge, MA USA
Locations (15):
- India (7):
  - Research Sites, Bangalore
  - Research Site, Chennai
  - Research Site, Hyderabaad
  - Research Site, Ludhiana
  - Research Site, Mumbai
  - Research Site, New Delhi
  - Research Site, Secunderabad
- Israel (4):
  - Research Site, Ashkelon
  - Research Site, Jerusalem
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- United Kingdom (4):
  - Research Site, Cambridge
  - Research Site, Manchester
  - Research Site, Norwich
  - Research Site, Salford